CLINICAL TRIAL: NCT00940069
Title: A Multicenter, Open Clinical Trial of Using TS Gene Polymorphism to Predict Effect in Patients of Advanced Lung Adenocarcinoma to Pemetrexed Combining With Cisplatin Regiment as First-line Treatment
Brief Title: TS Gene Polymorphism Predicts Effect in Patients With Advanced Lung Cancer
Acronym: TPEIAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yi Luo, director, Hunan Province Tumor Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LYN-LC-001
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Non-small-cell Lung Cancer; Adenocarcinoma
Keywords: TS; polymorphism; lung cancer; adenocarcinoma; pemetrexed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Lung Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TS high expression genotype (Experimental): TS high expression genotype delivered to pemetrexed 500 mg/m2 and cisplatin 75 mg/m2,for not less than 4 cycle, administered intravenously every 3 weeks.
  Interventions: Drug: pemetrexed
- TS low expression genotype (Experimental): TS low expression genotype delivered to pemetrexed 500 mg/m2 and cisplatin 75 mg/m2,for not less than 4 cycle, administered intravenously every 3 weeks.
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — 'TS high expression genotype': pemetrexed 500 mg/m2 and cisplatin 75 mg/m2 on day 1 of each 21 day,for not less than 4 cycle, administered intravenously every 3 weeks.
  'TS low expression genotype': pemetrexed 500 mg/m2 and cisplatin 75 mg/m2 on day 1 of each 21 day,for not less than 4 cycle, administered intravenously every 3 weeks.
  Other Names: Alimta

SUMMARY:
The investigators performed a multicenter, open trial of using TS gene polymorphism to predict advanced lung adenocarcinoma effect to pemetrexed combined with cisplatin regiment as first-line treatment.

DETAILED DESCRIPTION:
1. Main eligibility criteria were histologic or cytologic proof of advanced non-small-cell lung cancer (NSCLC) primary treatment, normal organ function, and Eastern Cooperative Oncology Group performance status 0 to 2.
2. All Patients were delivered to pemetrexed 500 mg/m2 and cisplatin 75 mg/m2 for not less than 4 cycle, administered intravenously every 3 weeks. Response assessment was performed every 6 weeks; toxicity assessment was performed every 3 weeks.
3. Primary end point was time to progression (TTP); secondary end points were objective response rate (ORR), overall survival (OS), and toxicity.
4. The study was designed to evaluate TS(thymidylate synthase) gene polymorphism as a predictor for advanced lung adenocarcinoma effect to pemetrexed combined with cisplatin regiment as first-line treatment.
5. Polymorphisms of thymidylate synthase were investigated in peripheral WBC（white blood cell）of all patients.

ELIGIBILITY:
Inclusion Criteria:

* histologic or cytologic proof of advanced lung adenocarcinoma
* primary treatment
* normal organ function
* Eastern Cooperative Oncology Group performance status 0 to 2

Exclusion Criteria:

* Symptomatic patients with brain metastases
* Major organ dysfunction and severe heart disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2013-06 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
time to progress | 6 months

SECONDARY OUTCOMES:
overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yi Luo, doctor, Study Chair — Hunan Province Tumor Hospital; Nong Yang, doctor, Principal Investigator — Hunan Province Tumor Hospital
Locations (1):
- HuNan province tumor hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Krawczyk P, Kucharczyk T, Kowalski DM, Powrozek T, Ramlau R, Kalinka-Warzocha E, Winiarczyk K, Knetki-Wroblewska M, Wojas-Krawczyk K, Kalakucka K, Dyszkiewicz W, Krzakowski M, Milanowski J. Polymorphisms in TS, MTHFR and ERCC1 genes as predictive markers in first-line platinum and pemetrexed therapy in NSCLC patients. J Cancer Res Clin Oncol. 2014 Dec;140(12):2047-57. doi: 10.1007/s00432-014-1756-6. Epub 2014 Jul 16. PMID 25028118
- [Result] Wang X, Wang Y, Wang Y, Cheng J, Wang Y, Ha M. Association of thymidylate synthase gene 3'-untranslated region polymorphism with sensitivity of non-small cell lung cancer to pemetrexed treatment: TS gene polymorphism and pemetrexed sensitivity in NSCLC. J Biomed Sci. 2013 Jan 25;20(1):5. doi: 10.1186/1423-0127-20-5. PMID 23350714